CLINICAL TRIAL: NCT02309762
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single-Ascending Intravenous Doses of FB825
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of FB825 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fountain Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FB825CLCT01
Record Dates: First submitted 2014-11-14; First posted 2014-12-05 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FB825 (Experimental): 6 cohorts of subjects are planned to be dosed by IV injection, with single- ascending doses ranging from 0.003 - 10 mg/kg
  Interventions: Drug: FB825
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FB825 — FB825 will be supplied at a concentration of 20 mg/mL for a single dose IV injection
  Arms: FB825
Drug: Placebo — Solution containing no active ingredients
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of single-ascending IV doses of FB825

ELIGIBILITY:
Inclusion Criteria:

1. The subject is male or female between 18 and 55 years of age, inclusive.
2. All female subjects must have a negative serum pregnancy test at screening and on Day -1.
3. The subject has a body weight ≥50 kg at screening and a body mass index of 18 to 30 kg/m2, inclusive.
4. The subject has a good health condition based upon the results of medical history, physical examination, vital signs, laboratory profile and ECG.
5. The subject has a negative urine drug screen for alcohol, cotinine.

Exclusion Criteria:

1. Female subjects who are pregnant or lactating.
2. The subject has a past history of heart arrhythmias.
3. The subject has history of clinically significant diseases.
4. The subject has any history of a previous anaphylactic reaction.
5. Use of prescribed medication within 6 months of Day -1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse events (AE) | Up to day140
Clinical laboratory test results (hematology, coagulation, serum chemistry[including liver function tests], and urinalysis) | Up to day140
Vital sign measurements (systolic and diastolic blood pressures, heart rate, respiratory rate, and oral body temperature) | Up to day140
12-lead ECG results | Up to day140
Physical examination findings | Up to day140

SECONDARY OUTCOMES:
Composite of PK parameters | Pre-dose, 2, 3, 5, 14, 29, 85, and 140 day post-dose
  Blood will be collected for the determination of serum FB825 concentrations, Cmax, Tmax, AUC, and terminal half-life.These parameters will be determined using non-compartmental methods.
Total IgE serum concentrations | pre-dose, 5, 14, 29, 85, and 140 day post-dose
  Blood will be collected to measure serum IgE concentrations.
Immunogenicity (Anti-FB825 antibody in serum) | pre-dose, 5, 14, 29, 85, and 140 day post-dose
  Blood will be collected to measure Immunogenicity.